CLINICAL TRIAL: NCT02953093
Title: Study of Changes in Muscle and Fat Gene Transcription With Acarbose Treatment: a Crossover Study
Brief Title: Study of Acarbose in Longevity
Acronym: SAIL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Upon review it was determined that the study terminated early due to lack of funding. Study never reached enrollment target and was administratively closed out by the Albert Einstein College of Medicine IRB.
Sponsor: Montefiore Medical Center (Other)
Collaborators: Glenn Foundation for Medical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-6933
Record Dates: First submitted 2016-09-09; First posted 2016-11-02 (Estimated); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Aging
Keywords: acarbose; aging
MeSH Terms: interventions — Acarbose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acarbose first (Other): Participants will take acarbose three times daily for 10 weeks (titration over 4 weeks, maintenance 6 weeks). After a two week washout, participants will take placebo three times daily for a total of 10 weeks (titration over 4 weeks, maintenance 6 weeks).
  Interventions: Drug: Acarbose; Other: Placebo
- Placebo first (Other): Participants will take placebo three times daily for 10 weeks (titration over 4 weeks, maintenance 6 weeks). After a two week washout, participants will take acarbose three times daily for a total of 10 weeks (titration over 4 weeks, maintenance 6 weeks).
  Interventions: Drug: Acarbose; Other: Placebo

INTERVENTIONS:
Drug: Acarbose — see arm description
  Other Names: Precose
Other: Placebo — See arm description

SUMMARY:
The investigators are studying the effects of acarbose on muscle and adipose gene transcription in older adults.

DETAILED DESCRIPTION:
Acarbose, an FDA approved drug for the treatment of type 2 diabetes, has known effects on glucose metabolism. Evidence from mice indicates that acarbose may prolong lifespan. In humans, acarbose improves inflammatory markers and reduces cardiovascular events. Consequently, acarbose is of interest in clinical translational aging research since it may influence fundamental processes that contribute to age-related diseases. The study described herein is an exploratory study to examine the effect of acarbose treatment on the biology of aging in humans. Specifically, the investigators plan to study whether treatment with a 10 week course of acarbose will alter the gene expression profile in adipose tissue and muscle in older adults in pathways that are known to be affected by human aging, in a placebo-controlled crossover study.

ELIGIBILITY:
Inclusion Criteria:

* Male
* age >60 years
* impaired fasting glucose (IFG) or impaired glucose tolerance (IGT)

Exclusion Criteria:

* cancer
* heart failure
* Chronic Obstructive Pulmonary Disease (COPD)
* inflammatory conditions
* estimated Glomerular Filtration Rate (eGFR) <45
* active liver disease
* poorly controlled hypertension
* epilepsy
* recent cardiovascular disease event (last 6 months)
* inflammatory bowel disease
* history of bariatric or other gastric surgery
* cigarette smoking
* serious substance abuse.
* Treatment with drugs known to influence glucose metabolism
* Hypersensitivity to acarbose or any component of the formulation.
* Treatment with anti-coagulant medications or anti-platelet drugs

Ages: 60 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nir F Barzilai, MD, Principal Investigator — Albert Einstein College of Medicine Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to researchers who are not part of the study

RESULTS

PARTICIPANT FLOW:
Groups:
- Acarbose First, Then Placebo: Participants will take Acarbose three times daily for 10 weeks (titration over 4 weeks, maintenance 6 weeks as per protocol). After a two week washout period, participants will take Placebo three times daily for a total of 10 weeks (titration over 4 weeks, maintenance 6 weeks as per protocol).
- Placebo First, Then Acarbose: Participants will take Placebo three times daily for 10 weeks (titration over 4 weeks, maintenance 6 weeks as per Protocol). After a two week washout period, participants will take Acarbose three times daily for a total of 10 weeks (titration over 4 weeks, maintenance 6 weeks as per Protocol).
Period: First Intervention (10 Weeks)
Arm/Group | Acarbose First, Then Placebo | Placebo First, Then Acarbose
Started | 14 | 14
Completed | 10 | 10
Not Completed | 4 | 4
Period: Washout Period (2 Weeks)
Arm/Group | Acarbose First, Then Placebo | Placebo First, Then Acarbose
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention (10 Weeks)
Arm/Group | Acarbose First, Then Placebo | Placebo First, Then Acarbose
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acarbose First, Then Placebo | Placebo First, Then Acarbose | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Customized [Count of Participants; unit: Participants] — Age was presented using a customized format based on the eligibility criteria and cohort associated with the study.
  Participants
    60-81 years old | 10 | 10 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Tissue Gene Expression Using RNA Sequencing (RNA-Seq)
Description: Difference in gene expression in muscle and abdominal adipose tissue using RNA-Seq were to have been evaluated to assess the effects of absorbed metabolites on tissues. Muscle and adipose are key metabolic tissues that undergo significant age-related changes and play an active role in the pathogenesis of aging. Muscle and abdominal adipose tissue samples were obtained and homogenized with tissue homogenizer. Subsequent mRNA extraction and analysis of gene expression (RNA seq) was conducted using multiplexed 100bp single-end sequencing. Differential expression between samples and after acarbose and after placebo were to have been determined using a negative binomial model approach implemented in the DESeq package. Results were to have been summarized by study arm and subsequently analyzed.
Time Frame: 10 weeks
Population: Muscle and abdominal adipose tissue biopsies collected and processed for gene expression data analyses did not yield meaningful data as the results were unable to be differentially expressed and could not be reported. Funding for repeat assays was unavailable and this study was terminated and unable to be published. Funding required to repeat gene expression data analyses is not available and results for this Outcome Measure will never be able to be reported.
Arm/Group | Acarbose First, Then Placebo | Placebo First, Then Acarbose
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Serum microRNA (miRNA)
Description: Differences in miRNA expression between acarbose and placebo arms were to have been evaluated. 1 milliliter (mL) of sera collected from the processing of blood samples will be used for miRNA sequencing. miRNA was extracted from the serum samples using miRNeasy kit in accordance with the manufacturer's protocol and miRNA libraries were prepared. Cel-miR-39 mimic was added to each sample before extraction, for normalization, and sequenced using multiplexed single-end sequencing on an Illumina HiSeq2500. miRNA are small, non-coding RNAs that regulate gene expression at a post-transcriptional level. Due to their stability in blood, changes in expression of circulating miRNA may serve as markers for age-related pathologies and investigators have correlated B-lymphocyte miRNA profiles in the plasma associated with exceptional longevity. Read counts were to have been summarized by study arm and statistically analyzed using a Wilcoxon test to compare miRNA expression levels.
Time Frame: At the end of 10 week treatment period (Visit 4) and at 22 weeks (Visit 6) following enrollment
Population: Serum samples collected and pre-processed for microRNA expression level determinations were never sequenced and analyzed due to lack of funding. Since samples were never sequenced and analyzed there is no read count data to summarize and there are no results to report. Funding to sequence samples for analysis is not available and results for this Outcome Measure will never be able to be reported.
Arm/Group | Acarbose First, Then Placebo | Placebo First, Then Acarbose
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Fecal Microbiome for 16s Ribosomal DNA (rDNA) Gene Sequencing
Description: 16s rDNA gene sequence expression levels were to have been assessed following the collection of stool samples. A fecal microbiome stool collection kit was provided to participants for self-collection of samples and returned for treatment and analysis. 16s rDNA sequencing was to have been performed to assess bacterial species clustering. Fecal microbial DNA was extracted from the samples and eluted DNA divided into 1 cubic centimeter (cc) aliquots and shipped for 16s rDNA sequencing. The raw 16s sequence data was converted to taxonomic profiles by grouping 16s sequences into Operational Taxonomic Units (OTUs) based on sequence similarity as well as by generating de-novo OTU generation using a de novo OTU-picking tool. A Basic Local Alignment Search Tool (BLAST) was to have been used to analyze each OTU's representative against a database. Relative abundance plots for visual comparison of microbial abundances were to have been generated, summarized, and reported by study arm.
Time Frame: At the end of 10 week treatment period (Visit 4) and at 22 weeks (Visit 6) following enrollment
Population: Stool samples collected for 16S fecal microbiome analysis were submitted to an external laboratory for processing and analysis; however, results were confounding and uninterpretable. As such, relative abundance plots were unable to be generated. In the absence of relative abundance plots there is no gene expression data to review, summarize, or report. Funding required to repeat fecal microbiome analyses is not available and results for this Outcome Measure will never be able to be reported.
Arm/Group | Acarbose First, Then Placebo | Placebo First, Then Acarbose
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to the time of Visit 5 at 16 weeks, approximately 4 months total
Groups:
- Acarbose: Participants will take Acarbose three times daily for 10 weeks (titration over 4 weeks, maintenance 6 weeks as per protocol) either prior to their Placebo regimen or following their Placebo regimen, after a 2-week washout period.
- Placebo: Participants will take Placebo three times daily for 10 weeks (titration over 4 weeks, maintenance 6 weeks as per Protocol) either prior to their Acarbose regimen or following their Acarbose regimen, after a 2-week washout period.
Arm/Group | Acarbose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 3/20 | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acarbose (N=20) | Placebo (N=20)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Respiratory Tract Neoplasms
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acarbose (N=20) | Placebo (N=20)
Left Arm Discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 — Verbatim Term
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 — Verbatim Term
Gout Flare up (Musculoskeletal and connective tissue disorders) | 1 | 0 — Verbatim Term
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 — Verbatim Term
Flatulence (Increased) (Gastrointestinal disorders) | 1 | 0 — Verbatim Term
Mild Fibrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 — Verbatim Term: Mild Fibrosis in left periumbilical area
Hematoma (Vascular disorders) | 0 | 1 — Verbatim Term: Hematoma in left leg post-biopsy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT02953093/Prot_SAP_002.pdf
  • Informed Consent Form (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT02953093/ICF_001.pdf